CLINICAL TRIAL: NCT03837132
Title: The Impact of Early Palliative Care on the Quality of Life of Patients With Advanced Pancreas Cancer: A Case-crossover Study
Brief Title: Early Palliative Care on Quality of Life of Patients With Advanced Pancreas Cancer
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: CancerCare Manitoba (Other); Celgene (Industry)
Responsible Party: Principal Investigator, Christina Kim, Medical Oncologist, CancerCare Manitoba; Assistant Professor, University of Manitoba, University of Manitoba
Other Study IDs: H2018:291
Record Dates: First submitted 2018-08-08; First posted 2019-02-11 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Advanced Cancer
Keywords: Advanced Pancreatic Cancer; Early Palliative Care; Quality of Life

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced pancreatic cancers: Newly diagnosed patients with advanced pancreatic cancer
  Interventions: Behavioral: Palliative care assessment

INTERVENTIONS:
Behavioral: Palliative care assessment — Patients with advanced pancreatic cancer will have regular palliative care assessment with palliative care team
  Other Names: Early palliative care assessment

SUMMARY:
The primary objective is to explore the impact of early palliative care on quality of life in patients with advanced pancreatic cancer. The secondary objectives are to explore the impact of early palliative care on symptom management, depression, anxiety and survival in patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
This is a prospective case-crossover study of patients with advanced pancreatic cancer (APC) at CancerCare Manitoba (CCMB) with early palliative care (PALC) plus standard oncologic care.

The primary endpoint of this study is quality of life (QOL) at week 16, measured by the Functional Assessment of Cancer Therapy - hepatobiliary (FACT-Hep). FACT-hep is a 45-item tool, which measures physical, emotional, social and functional well-being, and has been validated in a general population with hepatobiliary cancers, including metastatic pancreatic cancer. FACT-Hep has strong psychometric properties, and is a reliable, comprehensive and well-validated scale for use in patients with gastrointestinal cancers.

Secondary endpoints will include: (1) symptom control at 16 weeks as measured by the revised Edmonton Symptom Assessment Scale (ESAS-r), (a widely used and validated tool to assess symptom intensity, which is routinely completed by patients at all CCMB visits); (2) depression and anxiety at 16 weeks using the Hospital Anxiety and Depression Scale (HADS), (a-14 item scale which can be used in the outpatient setting to screen for anxiety and depression within the previous week) and the Patient Health Questionnaire (PHQ-9), (a sensitive (88%) and specific (88%) 9-question tool which incorporates diagnostic criteria for major depression); and overall survival measured from date of registration to death.

Recruitment to the study will occur in a clinic staffed by medical oncologists with expertise in gastrointestinal cancers, as this is the first point of entry into the CCMB system for patients with APC.

Early PALC will consist of referral to PALC at the time of study enrollment. Patients will undergo an initial consultation by the PALC team within two weeks of registration. Patients enrolled in the study who are also receiving chemotherapy must have their initial PALC consultation before receiving cycle 2 of chemotherapy. Baseline QoL questionnaires may be completed any time between registration and the first PALC consultation. The PALC team will be led by a physician with subspecialty training in PALC and an advanced practice nurse, with the ability to involve other members of the team (dietician, pharmacist, social worker, psychologist, psychiatrist, spiritual care, home care) as needed. The initial consultation by the PALC team will consist of assessments as per guidelines set by the Canadian Hospice Palliative Care Association. Patients will be followed by the PALC team at least every 2 weeks for the first month, then every 4 weeks until week 16, then at the discretion of the PALC team thereafter. Follow-up PALC visits will occur in person or via telehealth videoconference. A more intensive follow up regimen will occur early on, with a goal of achieving symptom control, as APC related symptoms can result in emergency room visits and hospitalizations. Patients will also receive regular oncologic follow up as directed by their oncologist.

All patients will complete the FACT-hep, ESAS-r, HADS and PHQ-9 at baseline and every 4 weeks until week 16. The data collected at these time points will provide a sense of the trajectory of the patient experience and provide insights into the timing of interventions to improve management of pain, symptoms, anxiety and depression in the future. Measuring QOL at these various time points may also be useful in case we experience unexpected loss to follow up at weeks 16, as it would provide data at intermediate time points for analysis.

Completion of QOL questionnaires will take patients approximately 15-20 minutes (10-15 minutes for FACT-hep), 1-2 minutes for ESAS, 2-3 minutes for HADS, and 1-2 minutes for PHQ-9). Questionnaires will be completed in the outpatient clinic, at least 7 days after receiving any chemotherapy to avoid conflation from chemotherapy side effects. All questionnaires will be collected by a study coordinator, and the study coordinator will be available to assist patients with questionnaire paperwork as needed. If a patient does not have an oncology appointment, they may receive the questionnaires and a stamped return envelope in the mail. If the questionnaires are not returned within 2 weeks, the study coordinator will contact the patient via phone as a reminder. If necessary, the study coordinator can complete these in an interview-style format over the telephone.

Patient and treatment characteristics will be captured at baseline, including: age, sex, education level, height, weight, primary language spoken, Eastern Cooperative Oncology Group (ECOG) performance status, comorbid illnesses (hypertension, dyslipidemia, diabetes, coronary artery disease, cerebrovascular accident or transient ischemic attack, psychiatric illness, other cancers), medications (prescribed, over the counter, alternative/complementary), use of opioids for cancer related pain, weight loss, clinical stage (locally advanced, unresectable/metastatic), site of primary tumour in pancreas (head or neck/body/tail), CA 19-9 (normal/elevated). Emergency room visits and hospitalizations while on study will be captured. This data will be used to describe the study cohort. Data will be entered and maintained in REDCap on the University of Manitoba's secure research environment.

Note: During the time of the COVID-19 response, patients are assessed over the phone by the advanced practice nurse two days before their scheduled appointment to determine if in-person visits are necessary. If in-person visits are necessary, follow up palliative care visits will be done in clinic with only one support person allowed per patient and clinic visit time limited to minimize any potential exposure time. In in-person visits not necessary, the follow up palliative care visits are conducted over the phone until COVID-19 precautions are lifted.

ELIGIBILITY:
Inclusion Criteria:

* age >18
* newly diagnosed advanced pancreatic cancer (APC)
* English speaking or willing to be seen with a medical interpreter
* willing and able to complete quality of life (QoL) questionnaires

Exclusion Criteria:

* age <18
* receiving cycle 2 of chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed advanced adult pancreatic patients
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Impact of early palliative care on quality of life in patients with advanced pancreatic cancer | registration to 16 weeks
  For the primary endpoint, we will use a generalized linear model to test for a statistically significant change score between baseline and 16 weeks. We will assume a normal distribution for the change scores. Model fit will be assessed via a visual assessment of residuals and the ratio of the model deviance to its degrees of freedom.

SECONDARY OUTCOMES:
To explore the impact of early palliative care on symptom management, depression, anxiety and survival in patients with advanced pancreatic cancer | registration to 16 weeks
  Secondary endpoints will include: (1) symptom control at 16 weeks as measured by the revised Edmonton Symptom Assessment Scale (ESAS-r) (a widely used and validated tool to assess symptom intensity, which is routinely completed by patients at all CCMB visits); (2) depression and anxiety at 16 weeks using the Hospital Anxiety and Depression Scale (HADS) (a 14 item scale which can be used in the outpatient setting to screen for anxiety and depression within the previous week) and the Patient Health Questionnaire (PHQ-9) (a sensitive (88%) and specific (88%) 9 question tool which incorporates diagnostic criteria for major depression); and overall survival measured from date of registration to death

CONTACTS AND LOCATIONS:
Overall Officials: Christina Kim, MD FRCPC, Principal Investigator — CancerCare Manitoba/ University of Manitoba
Locations (1):
- Victoria General Hospital Buhler Cancer Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim CA, Lelond S, Daeninck PJ, Rabbani R, Lix L, McClement S, Chochinov HM, Goldenberg BA. The impact of early palliative care on the quality of life of patients with advanced pancreatic cancer: The IMPERATIVE case-crossover study. Support Care Cancer. 2023 Apr 6;31(4):250. doi: 10.1007/s00520-023-07709-3. PMID 37022483